CLINICAL TRIAL: NCT02720315
Title: Intensive Cryotherapy in the Emergency Department (ICED) Versus Conventional Treatment for Acute Musculoskeletal Injuries: The ICED Randomized Controlled Trial
Brief Title: Intensive Cryotherapy in the Emergency Department for Acute Musculoskeletal Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Eric Leroux, Chief Resident, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 34835
Record Dates: First submitted 2016-03-10; First posted 2016-03-25 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Pain; Opiate; Emergency
MeSH Terms: conditions — Pain; Emergencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive cryotherapy (Experimental): Application of ice in a plastic bag wrapped to the patient's site of pain, and kept in place for 20min.
  Interventions: Procedure: Intensive cryotherapy
- Control (No Intervention): Existing pain control practice of physicians and nurses, which includes application of a chemical cold pack.

INTERVENTIONS:
Procedure: Intensive cryotherapy — Application of ice inside a plastic bag wrapped to the patient's site of pain, and held in place for 20min.
  Arms: Intensive cryotherapy

SUMMARY:
Acute musculoskeletal (MSK) injuries, including strains, sprains or contusions, are a common reason patients seek emergency care. Pain control is an essential component of treatment. Within the orthopedic literature, there is robust body of research supporting the use of cryotherapy for post-operative patients and injured athletes. However, within the emergency department (ED), studies have been focused on pharmacologic analgesia. The absence of evidence on optimal method or impact of ice therapy for acute MSK injuries contributes to inconsistent practice patterns that may impede symptom control or increase narcotic usage.

The specific aim of the ICED investigation is to evaluate the effectiveness of intensive cryotherapy for the treatment of pain due to acute MSK injuries treated in the ED. Secondary outcomes include length-of-stay (LOS), patient satisfaction, and narcotic usage.

DETAILED DESCRIPTION:
Background Acute musculoskeletal (MSK) injuries, including strains, sprains or contusions, are a common reason patients seek emergency care. Pain control is an essential component of treatment. Within the orthopedic literature, there is robust body of research supporting the use of cryotherapy for post-operative patients and injured athletes. However, within the emergency department (ED), studies have been focused on pharmacologic analgesia. The absence of evidence on optimal method or impact of ice therapy for acute MSK injuries contributes to inconsistent practice patterns that may impede symptom control or increase narcotic usage.

Objectives The specific aim of the ICED investigation is to evaluate the effectiveness of intensive cryotherapy for the treatment of pain due to acute MSK injuries treated in the ED. Secondary outcomes include length-of-stay (LOS), and narcotic usage.

Methods Adults younger than sixty-six years-old presenting to the ED with acute MSK pain are enrolled through a process of informed consent, unless one or more of the exclusion criteria are met. Crushed ice is double-bagged and applied at the site of injury, where it is wrapped in place for twenty minutes. Pain scores are measured using a visual analog scale (VAS) when the ice is applied, at 20 minutes and at 60 minutes. Treating physicians do not alter their management. Data on LOS and use of pharmacologic analgesics are obtained through chart review.

Results Change in VAS will be analyzed with regression analysis and analysis of variance. Patients are grouped into categories of pharmacologic analgesic usage. Patient satisfaction scores and narcotic usage will be analyzed using a Chi Square test, while LOS data compared with an unpaired two-tailed t-test.

ELIGIBILITY:
Inclusion Criteria:

* all people presenting to the ED with musculoskeletal injuries

Exclusion Criteria:

* Patients with hip fractures
* Patients with open fractures
* Patients with altered mental status who are unable to consent to participate in the study
* Patients activated as a trauma
* Patients with fractures or dislocations requiring closed reduction in the emergency department
* Minors
* Prisoners
* Patients with known pregnancy
* Patient who are receiving investigational drug as part of another study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Change in pain level | 20 minutes
Change in pain level | 60 minutes

SECONDARY OUTCOMES:
Change in analgesic utilization | 24hr
  Measured by chart review to detail the type and quantity of analgesics utilized by the control and the intervention groups.

IPD SHARING:
Plan to Share IPD: No